CLINICAL TRIAL: NCT01231698
Title: Strict Heart Rate Control With Esmolol in Septic Shock: a Randomized, Controlled, Clinical Pilot Study
Brief Title: Heart Rate Control With Esmolol in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea Morelli (Other)
Responsible Party: Sponsor-Investigator, Andrea Morelli, MD, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2048
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2011-11

CONDITIONS: Septic Shock
Keywords: septic shock; esmolol; tachycardia; betablockers
MeSH Terms: conditions — Shock, Septic; Tachycardia | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- esmolol (Experimental)
  Interventions: Drug: esmolol
- control (Other)
  Interventions: Other: control

INTERVENTIONS:
Drug: esmolol — Strict heart rate control: esmolol at any dose to maintain heart rate between 95 and 80 bpm.
  Arms: esmolol
Other: control — standard treatment without strict heart rate control
  Arms: control

SUMMARY:
The purpose of this study is investigate the effects on systemic hemodynamics and organ function of esmolol when used to maintain heart rate below a predefined threshold in patients with septic shock.

DETAILED DESCRIPTION:
154 septic shock patients with heart rate > of 95 bpm and requiring vasopressor support to maintain mean arterial pressure between 65 and 75 mmHg despite adequate volume resuscitation, will be enrolled in the study. Patients will be randomly allocated to be treated with either a) a continuous esmolol infusion at any doses to maintain heart rate between 95 and 80 bpm b)to a standard treatment without heart rate control(control; each n = 77). In both groups, norepinephrine will be titrated to achieve a mean arterial pressure (MAP) between 65 and 75 mmHg. Data from right heart catheterization,data from organ function as well as norepinephrine requirements will be obtained at baseline and after 24, 48, 72, and 96 hours. The protocol will require that esmolol be infused continuously at any doses to maintain the predefined heart rate threshold until one the following events occur: the patient die, a serious adverse effect attributed to the study drug infusion, or the patient has been discharged from ICU.

ELIGIBILITY:
Inclusion Criteria:

* septic shock criteria
* presence of heart rate > 95 bpm.

Exclusion Criteria:

* Pregnancy
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
heart rate | over a period of 96 hrs

SECONDARY OUTCOMES:
systemic hemodynamics | over a period of 96 hours
  systemic hemodynamics,norepinephrine requirements,organ functions,adverse effects.

OTHER OUTCOMES:
ICU Mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Anesthesiology and Intensive care of the University of Rome La Sapienza, Rome, Italy

REFERENCES:
- [Derived] Morelli A, Ertmer C, Westphal M, Rehberg S, Kampmeier T, Ligges S, Orecchioni A, D'Egidio A, D'Ippoliti F, Raffone C, Venditti M, Guarracino F, Girardis M, Tritapepe L, Pietropaoli P, Mebazaa A, Singer M. Effect of heart rate control with esmolol on hemodynamic and clinical outcomes in patients with septic shock: a randomized clinical trial. JAMA. 2013 Oct 23;310(16):1683-91. doi: 10.1001/jama.2013.278477. PMID 24108526